CLINICAL TRIAL: NCT03526055
Title: Evaluation of Clinical Outcomes of Pulse Widths <500 µS And >1000 µS During a Temporary Spinal Cord Stimulation Trial
Brief Title: Evaluation of Conventional and Long Pulse Widths During a Temporary Spinal Cord Stimulation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amol Soin (Other)
Responsible Party: Sponsor-Investigator, Amol Soin, Principal Investigator, Kettering Health Network
Organization: Kettering Health Network (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Long Pulse
Record Dates: First submitted 2018-03-06; First posted 2018-05-16 (Actual); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: Spinal Cord Stimulation; Pain, Back; Pain
MeSH Terms: conditions — Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- <500 µS Pulse Width (Active Comparator): Intervention includes spinal cord stimulation will be programmed to <500 µS pulse width and patient will undergo an Algovita Spinal Cord Stimulation System trial procedures. Following the trial procedure, the subject's EPG will be set to the appropriate pulse width, based on the arm assigned, and then programmed to achieve optimal pain relief.
  Interventions: Device: Algovita Spinal Cord Stimulation System
- >1000 µS Pulse Width (Experimental): Intervention includes spinal cord stimulation will be programmed to >1000 µS pulse width and patient will undergo an Algovita Spinal Cord Stimulation System trial procedures. Following the trial procedure, the subject's EPG will be set to the appropriate pulse width, based on the arm assigned, and then programmed to achieve optimal pain relief.
  Interventions: Device: Algovita Spinal Cord Stimulation System

INTERVENTIONS:
Device: Algovita Spinal Cord Stimulation System — The Algovita™ SCS system is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with failed back surgery syndrome, intractable low back pain and leg pain.

SUMMARY:
The purpose of this study is to evaluate the effect of pulse widths <500 µS and >1000 µS on clinical outcomes during a temporary SCS trial.

DETAILED DESCRIPTION:
The proposed study is a prospective, single-center, two arm, randomized, crossover design to be conducted at The Ohio Pain Clinic. The study will enroll up to 15 subjects in order to include up to 10 subjects in the study. Subjects selected to participate in the trial have back and/or leg pain, have been evaluated as a candidate for SCS and have agreed to undergo a temporary SCS trial using the Algostim system with percutaneous leads. Each subject will be followed during the trial period of approximately 7 days.

The study will end when the last subject has completed the trial period. exited. The expected enrollment period for this study is approximately three months. After exit from the clinical study, subjects will continue to be followed by their physician per usual care. All device and procedure-related AEs will be collected and reported per the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subject is eligible for SCS therapy according to the Algovita SCS system Indications for Use statement
* Study candidate is undergoing a SCS trial using Nuvectra Algostim system
* Subject signed a valid, Institutional Review Board (IRB)-approved informed consent form.
* Subject is 18 years of age or older when written informed consent is obtained

Exclusion Criteria:

* Subject is contraindicated for an Algovita SCS system
* Subject has a cognitive impairment or exhibits any characteristic, that would limit the study candidate's ability to assess pain relief or complete study assessments
* Subject has a life expectancy of less than 2 years
* Subject is participating in another clinical study that would confound data analysis
* Subject has a coexisting pain condition that might confound pain ratings
* Subject has a significant psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol Soin, MD, MBA, Principal Investigator — Ohio Pain Clinic
Locations (1):
- Ohio Pain Clinic, Centerville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Chronic Pain Association Resource Guide to Chronic Pain Medication and Treatment, 2014 Edition.
- [Background] North RB, Campbell JN, James CS, Conover-Walker MK, Wang H, Piantadosi S, Rybock JD, Long DM. Failed back surgery syndrome: 5-year follow-up in 102 patients undergoing repeated operation. Neurosurgery. 1991 May;28(5):685-90; discussion 690-1. PMID 1831546
- [Background] Wilkinson HA. The Failed Back Surgery Syndrome: Etiology and Therapy, 2nd edition., Philadelphia: Harper & Row, 1991.
- [Background] Law JD, Lehman RA, Kirsch WM. Reoperation after lumbar intervertebral disc surgery. J Neurosurg. 1978 Feb;48(2):259-63. doi: 10.3171/jns.1978.48.2.0259. PMID 146731
- [Background] Lehmann TR, LaRocca HS. Repeat lumbar surgery. A review of patients with failure from previous lumbar surgery treated by spinal canal exploration and lumbar spinal fusion. Spine (Phila Pa 1976). 1981 Nov-Dec;6(6):615-9. PMID 6461073
- [Background] Jobling DT, Tallis RC, Sedgwick EM, Illis LS. Electronic aspects of spinal-cord stimulation in multiple sclerosis. Med Biol Eng Comput. 1980 Jan;18(1):48-56. doi: 10.1007/BF02442479. No abstract available. PMID 6966725
- [Background] Davis R, Gray E. Technical factors important to dorsal column stimulation. Appl Neurophysiol. 1981;44(1-3):160-70. doi: 10.1159/000102196. PMID 6975071
- [Background] Holsheimer J. Effectiveness of spinal cord stimulation in the management of chronic pain: analysis of technical drawbacks and solutions. Neurosurgery. 1997 May;40(5):990-6; discussions 996-9. doi: 10.1097/0006123-199705000-00023. PMID 9149258
- [Background] Gould B, Bradley K. Pulse width programming in spinal cord stimulators. Abstract of the American Academy of Pain Medicine 22nd Annual Meeting, 2006 February 22-25. San Diego, CA
- [Background] Yearwood TL, Hershey B, Bradley K, Lee D. Pulse width programming in spinal cord stimulation: a clinical study. Pain Physician. 2010 Jul-Aug;13(4):321-35. PMID 20648201
- [Background] Lee D, Hershey B, Bradley K, Yearwood T. Predicted effects of pulse width programming in spinal cord stimulation: a mathematical modeling study. Med Biol Eng Comput. 2011 Jul;49(7):765-74. doi: 10.1007/s11517-011-0780-9. Epub 2011 Apr 29. PMID 21528381
- [Background] Grill WM Jr, Mortimer JT. The effect of stimulus pulse duration on selectivity of neural stimulation. IEEE Trans Biomed Eng. 1996 Feb;43(2):161-6. doi: 10.1109/10.481985. PMID 8682527

RESULTS

PARTICIPANT FLOW:
Groups:
- <500 µS Pulse Width First, Then >1000 µS Pulse Width: Intervention includes spinal cord stimulation will be programmed to <500 µS pulse width and patient will undergo an Algovita Spinal Cord Stimulation System trial procedures. Following the trial procedure, the subject's EPG will be set to the appropriate pulse width, based on the arm assigned, and then programmed to achieve optimal pain relief.
  Algovita Spinal Cord Stimulation System: The Algovita™ SCS system is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with failed back surgery syndrome, intractable low back pain and leg pain.
- >1000 µS Pulse Width First, Then <500 µS Pulse Width: Intervention includes spinal cord stimulation will be programmed to >1000 µS pulse width and patient will undergo an Algovita Spinal Cord Stimulation System trial procedures. Following the trial procedure, the subject's EPG will be set to the appropriate pulse width, based on the arm assigned, and then programmed to achieve optimal pain relief.
  Algovita Spinal Cord Stimulation System: The Algovita™ SCS system is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with failed back surgery syndrome, intractable low back pain and leg pain.
Period: Initial Program
Arm/Group | <500 µS Pulse Width First, Then >1000 µS Pulse Width | >1000 µS Pulse Width First, Then <500 µS Pulse Width
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Program
Arm/Group | <500 µS Pulse Width First, Then >1000 µS Pulse Width | >1000 µS Pulse Width First, Then <500 µS Pulse Width
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This information was not collected. Although the protocol states that demographic information would be collected at baseline, the sponsor ended up not collecting this information.
Groups:
- Entire Study Population: Crossover study design, all participant data is collected together.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subject Pain Relief
Description: The study used a pain relief scale (similar to a brief pain inventory). The scale assessed pain relief using a percent relief rating in 10% increments, where a higher number represents greater pain relief than a lower number for the pain scale. A higher number is considered better for pain relief scale. The scale range is from 0%, which is no relief of pain to 100%, which is complete relief of pain. Subjects are asked to rate their pain by marking the box beside the number that best describes their pain in the last 24 hours.
Time Frame: up to 8 days
Measure: Mean (Full Range); unit: percentage of pain relief
Arm/Group | <500 µS Pulse Width | >1000 µS Pulse Width
Number analyzed (Participants) | 10 | 10
percentage of pain relief | 56 [0 to 100] | 61 [30 to 90]

2. Secondary Outcome: Distribution of Paresthesia
Description: 1. At end of each arm, subjects will be asked to complete a diagram that shows distribution of paresthesia.
Time Frame: Up to 8 days
Population: This information was not collected.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 0

3. Secondary Outcome: Subject Preference
Description: Subjects will be asked to select their favorite program
Time Frame: Up to 8 days
Population: 1 subject preferred both programs equally.
Measure: Count of Participants; unit: Participants
Arm/Group | <500 µS Pulse Width | >1000 µS Pulse Width
Number analyzed (Participants) | 10 | 10
Participants | 4 | 7

4. Secondary Outcome: Quality of Pain Relief
Description: Subjects will be asked to rate the quality of the pain relief achieved during the trial (from either arm) using the following scale; Excellent, Very Good, Good, Fair or Poor
Time Frame: Up to 8 days
Population: This information was not collected.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 0

5. Secondary Outcome: Subject Satisfaction
Description: Subjects will be asked to rate their overall satisfaction with the pain relief achieved during the trial (from either arm) using the following scale; Very Satisfied, Satisfied, Neither Satisfied nor Unsatisfied, Unsatisfied or Very Unsatisfied
Time Frame: Up to 8 days
Population: This information was not collected.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 0

6. Secondary Outcome: Achievement of ≥50% Pain Relief
Description: Number of patients who achieved ≥ 50% pain relief during the trial (from either arm). The study used a pain relief scale (similar to a brief pain inventory). The scale assessed pain relief using a percent relief rating in 10% increments, where a higher number represents greater pain relief than a lower number for the pain scale. A higher number is considered better for pain relief scale.
Time Frame: Up to 8 days
Population: 10 patients in total, crossover design.
Measure: Count of Participants; unit: Participants
Arm/Group | <500 µS Pulse Width | >1000 µS Pulse Width
Number analyzed (Participants) | 10 | 10
Participants | 5 | 8

7. Secondary Outcome: Rate of AEs
Description: Rate of device-related and/or procedure-related AEs
Time Frame: From spinal cord stimulation implant through study completion or study exit, Up to 8 days
Population: 10 patients total, crossover design
Measure: Number; unit: participants experienced AE
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
participants experienced AE | 0

ADVERSE EVENTS:
Time Frame: Up to 8 days
Groups:
- <500 μS Pulse Width: Intervention includes spinal cord stimulation will be programmed to <500 µS pulse width and patient will undergo an Algovita Spinal Cord Stimulation System trial procedures. Following the trial procedure, the subject's EPG will be set to the appropriate pulse width, based on the arm assigned, and then programmed to achieve optimal pain relief.
- >1000 μS Pulse Width: Intervention includes spinal cord stimulation will be programmed to >1000 µS pulse width and patient will undergo an Algovita Spinal Cord Stimulation System trial procedures. Following the trial procedure, the subject's EPG will be set to the appropriate pulse width, based on the arm assigned, and then programmed to achieve optimal pain relief.
Arm/Group | <500 μS Pulse Width | >1000 μS Pulse Width
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT03526055/Prot_000.pdf